CLINICAL TRIAL: NCT07115017
Title: Investigation of Inflammation Using [18F]FZTA
Brief Title: This Study Involves a Positron Emission Tomography (PET) Scan Using a New Investigational Radioactive Tracer, [18F]-FZTA, to Detect Inflammation in the Brain. The Tracer Will be Tested in Healthy Younger Adults and Individuals With Multiple Sclerosis.
Acronym: FZTA Pilot
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Tammie L. S. Benzinger, MD, PhD, Hugh Monroe Wilson Professor of Radiology, Washington University School of Medicine
Other Study IDs: 202505042
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for future research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Healthy participants will receive a single intravenous bolus injection of 7 ± 20% milliCurie (mCi) of the investigational radiotracer [18F]-FZTA. Participants will then undergo [18F]-FZTA PET scan.
  Interventions: Drug: [18F] FZTA
- Participants with Multiple Sclerosis: Participants with Multiple Sclerosis will receive a single intravenous bolus injection of 7 ± 20% milliCurie (mCi) of the investigational radiotracer [18F]-FZTA. Participants will then undergo a brain [18F]-FZTA PET scan
  Interventions: Drug: [18F] FZTA

INTERVENTIONS:
Drug: [18F] FZTA — Participants will receive a single intravenous bolus injection of 7 ± 20% milliCurie (mCi) of the investigational radiotracer [18F]-FZTA. A PET-certified medical professional will prepare and administer the [18F]-FZTA. Prior to the administration, the dosage will be assayed in a dose calibrator and diluted with 0.9% sodium chloride (normal saline) up to a total 20 mL syringe volume. Participants will receive a maximum intravenous bolus injection of 7+20% mCi of [18F]-FZTA followed by a 10 mL 0.9% sodium chloride (normal saline) flush.

SUMMARY:
This study involves a Positron Emission Tomography (PET) scan using a new investigational radioactive tracer, [18F]-FZTA, to detect inflammation in the brain. The tracer will be tested in healthy younger adults and individuals with Multiple Sclerosis.

DETAILED DESCRIPTION:
The primary objective of this initial IND study is to evaluate the safety of [18F]-FZTA for PET imaging of S1P1 expression. The study will begin with whole-body PET dosimetry in healthy adult volunteers to determine the safety and safe radiation dose for a single PET scan in humans. Following this, brain and neck imaging will be conducted in both healthy adult control participants and individuals with multiple sclerosis (both male and female) to characterize [18F]-FZTA uptake in the brain. An analysis of the radiolabeled metabolite will also be completed as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any race
* Age ≥ 18 years
* Capable of providing written informed consent for volunteering to undergo research procedures.
* Healthy volunteer or volunteer with a diagnosis of MS established using the revised McDonald criteria (2017)

Exclusion Criteria:

* Hypersensitivity to [18F]FZTA or any of its excipients;
* Contraindications to PET, CT, or MRI (e.g., certain incompatible electronic medical devices, inability to lie still for extended periods) that make it potentially unsafe for the individual to participate.
* Severe claustrophobia
* Women who are currently pregnant or breastfeeding
* Currently undergoing radiation therapy
* Any condition that, in the opinion of the Sponsor-Investigator or designee could increase risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection of the data (e.g., renal or liver failure, advanced cancer);
* Participants who in the last 6 months experienced any of the following cardiovascular conditions or findings in the screening electrocardiogram (ECG): clinically significant cardiac arrhythmias including atrial fibrillation with rapid ventricular response, myocardial infarction, high-grade heart block (type 2 or greater), unstable angina, stroke, transient ischemic attack or decompensated heart failure requiring hospitalization or Class III/IV heart failure;
* Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aim 1: Dosimetry/Safety group will consist of 10 healthy adult normal volunteers (5 males and 5 females) who will be recruited and undergo whole-body PET/CT imaging to assess the safety, dosimetry, and metabolism of [F-18]FZTA. All 10 participants will also undergo a short MRI without contrast.
  Aim 2: Proof of Concept/Healthy Cohort will consist of 15 healthy adult volunteers (Males and Females).
  Aim 3: Proof of Concept/MS cohort consists of 10 MS patients who are on stable therapy.
  Aim 4: Proof of Concept/MS cohort consists of newly diagnosed 20 RRMS patients who will be started on high-efficacy drugs.
  Aims 2,3, and 4 will undergo [F-18]FZTA PET imaging of the brain and neck, brain MRI, and an optional [C-11]CS1P1 and [F-18]FDG PET imaging.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
PET imaging studies of [18F]-FZTA in healthy control participants and participants with Multiple Sclerosis, and measuring the uptake of [18F]-FZTA tracer. | Through study completion, an average of 2 years
  To test the hypothesis that specific binding of [18F]-FZTA is elevated in participants with Multiple Sclerosis compared to healthy normal control participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD., PhD., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States